CLINICAL TRIAL: NCT06986772
Title: [14C]TGRX-678 Mass Balance Study in Chinese Healthy Male Adults
Brief Title: TGRX-678 Pharmacokinetic Mass Balance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-678-1003
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TGRX-678 (Experimental): healthy male subjects will be given 240mg/250uCi[14C]TGRX-678 in suspension
  Interventions: Drug: [14C]TGRX-678

INTERVENTIONS:
Drug: [14C]TGRX-678 — Healthy subjects will be given TGRX-678 240 mg orally on day 1.

SUMMARY:
This is a pharmacokinetic study for [14C]TGRX-678 on mass balance to evaluate distribution, metabolism and excretion of TGRX-678, a tyrosine kinase inhibitor indicated for treatment of chronic myeloid leukemia.

DETAILED DESCRIPTION:
This study is designed as a single-center, single-dose, non-randomized and open-label study. The study will be conducted in healthy male participants to evaluate distribution, metabolic pathways and route of excretion of TGRX-678 using the Carbon-14 labelled isotope of TGRX-678 compound. Safety and pharmacokinetic evaluation will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* age between 18 and 45 (both included) years old
* body weight index between 19.0 and 26.0 kg/m2 (both included, and body weight not lower than 50 kg
* can volunteeringly consent
* can communicate well with investigators and complete study according to protocol requirements

Exclusion Criteria:

* abnormal and of clinical significance results on physical exam, regular laboratory tests, thyroid function, anal check, chest x-ray, abdominal ultrasound check or 12-lead ECG
* positive test results on hepatitis B surface antigen/ E antigen, hepatitis C antibody, HIV antigen/antibody or syphylus antibody
* abnornal and of clinical significance results on eye exam
* usage of any inducers or inhibitors for drug metabolism enzymes (especially CYP3A4) within 30 days of screening
* usage of any prescriptional drug, OTC drug, herbal medicine, traditional Chinese medicine, or food supplements (i.e., vitamins, calcium) within 14 days of screening
* history of any clinically significant serious diseases or any conditions that at investigator's discretion may affect study results
* have condition that may affect drug absoption
* received major surgery or with un-healed surgical wounds within 6 months of screening
* have allergies to at least 2 substances or at investigator's discretion may be allergic to investigational drug or any excipients
* have hemorrhoids; have history of or is having conditions that cause bloody feces, irritable bowel syndrome, or inflammatory bowel disease
* habitutory constipation or diarrhea
* alcohol abuse, or frequent use of alcohol within 6 months of screening
* smoking of more than 5 cigarettes per day within 3 months of screening, or habitutory use of nicotine products and cannot quit during study
* drug abuse, or use of soft drug (marajuana) within 3 months of screening, or use of hard drug (phenylamine or PCP type drugs) within 1 year of screening, or tested positive in urine drug test during screening
* habitutory use of grape fruit juice, or overuse of tea, coffee or caffeinated drugs, and cannot quit during study
* long-term occupational exposure to radioactive conditions, or have history of significant radioactive substance exposure or participated in clinical study using radioactive-labeled drugs within 1 year of current study
* Having difficulties to receive venous needle puncture, or cannot tolerate venous needle puncture, or history of hematophobia or needle sickness
* Participation in any other clinical studies within 3 months before screening
* Reception of vaccine within 1 months before screening, or planning to be vaccinated during the study
* Planning to have children or donate sperms during the study and within 1 year after the study, or Not agreeing to take contraceptive measures during and within 1 year after study completion
* Blood donation or blood loss of > 400 ml within 3 months before screening; blood donation or blood loss of > 200 ml within 1 month before screening; reception of blood transfusion within 1 months before screening; received blood donation within 1 months of study, or planning to donate blood within 3 months after study completion
* Having special dietary requirements and unable to follow the uniform dietary plan in the study
* Any conditions that the investigator deemed unfit for the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Urine radioactivity | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  [C14]TGRX-678 radioactivity detected in urine
Fecal radioactivity | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  [C14]TGRX-678 radioactivity detected in feces
Plasma AUC (Area under curve) percentage | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  percentage of [C14]TGRX-678 radioactivity in plasma
Urine %Dose | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  percentage of [C14]TGRX-678 radioactivity in urine
Fecal %Dose | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  percentage of [C14]TGRX-678 radioactivity in feces
Plasma Cmax | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  Maximum concentration of [C14]TGRX-678 measured in plasma
Plasma Tmax | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  Time to maximum concentration of [C14]TGRX-678 measured in plasma
Plasma AUC(0-t) | Day-1 (day before dosing), Day 1 to Day 54 after dosing
  Area under curve for TGRX-678 plasma concentration from before dose to last measureable timepoint

SECONDARY OUTCOMES:
Adverse events/serious adverse events | Day-1 (day before dosing), Day 1 to Day 54 after dosing or the day sample collection is completed
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No